CLINICAL TRIAL: NCT04684095
Title: The Effect of ePRO on Quality of Life and Prognosis of Patients With Unresectable Metastatic Colorectal Cancer Who Received Bevacizumab Combined With Chemotherapy for First Line Treatment
Brief Title: The Effect of ePRO on Quality of Life and Prognosis of Patients With Unresectable Metastatic Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yanqiao Zhang, Director of the hospital, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EPRO-CRCQoL-1L
Record Dates: First submitted 2020-12-09; First posted 2020-12-24 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Colorectal Cancer Metastatic; Cancer
Keywords: Patient-Reported Outcomes; QoL; mCRC; Bevacizumab
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine follow-up group (No Intervention): only according to the routine follow-up frequency to the center visit.
- ePRO group (Experimental): ePRO group : self-evaluation in ePRO mode was accepted, and the patients were visited in the center according to the routine follow-up frequency.
  Interventions: Behavioral: electronic patient report outcome

INTERVENTIONS:
Behavioral: electronic patient report outcome — ePRO was conducted every two weeks in addition to routine follow-up
  Arms: ePRO group

SUMMARY:
Bevacizumab combined with fluorouracil-based chemotherapy is the first-line standard treatment for patients with metastatic colorectal cancer (mCRC). However, some research show that the long-term survival benefit of patients in real world data is inferior to clinical trial. The reason may be related to the difference in follow-up strategy of patients in the real world. Patient-Reported Outcomes (PROs) are a kind of outcome indicators that directly measure and evaluate the disease and its consequences based on how the patient feels about his own health. In advanced cancer, quality of life (QoL) is a major treatment goal. And the electronic patient report outcome (ePRO) has become an effective method to capture the symptoms of patients, which can improve the quality of life and physical and mental health of patients. In order to observe whether ePRO can bring clinical benefits to patients with metastatic colorectal cancer, this study aimed to compare the effects of ePRO and routine follow-up on the quality of life and prognosis of patients with unresectable metastatic colorectal cancer who received first-line bevacizumab combined with chemotherapy. This is an open label, multicenter, randomized controlled prospective study of first-line bevacizumab combined with chemotherapy in patients with unretractable metastatic colorectal cancer.The aim of this study was to assess the impact of ePRO on quality of life and survival outcomes compared with routine follow-up.The study intends to start in February 2021 and end in June 2024.Patients were recruited for 12 months and followed up for 24 months.The study included a screening period (28 days before first-line treatment to 1 day before treatment) and an observation period (from the beginning of treatment to the end of the study).Day 1 (baseline) was defined as the first day of first-line bevacizumab combined with chemotherapy.About 338 patients will be enrolled in the study in China, and enrolled patients will be randomly assigned to one of the following two groups in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have informed consent form (ICF) signed for the study
* Patients must be ≥18 years old when signing the ICF
* Histologically or cytologically-diagnosed unresectable metastatic colorectal cancer
* Patients must receive bevacizumab combined with chemotherapy for first-line systemic treatment
* The researcher believes that the patient is capable of implementing the research protocol

Exclusion Criteria:

* Patients has participated in any clinical trial in the past 4 weeks
* Patients is currently or about to participate in a clinical trial
* Patients with other malignant tumors (except carcinoma in situ)
* Patients with lung metastases only
* Patients with evidence of any serious or uncontrolled systemic disease, including but not limited to: unstable or decompensated respiratory, heart, liver or kidney disease, HIV infection, uncontrolled hypertension, diabetes, severe arrhythmia, massive hemorrhagic activity, etc
* Patients with history of alcohol or drug abuse
* According to the researcher's judgment, the possibility of inclusion is low (including inability to understand the study requirements, poor compliance, weakness, inability to ensure that the protocol can be implemented as required, etc.), or the researcher believes that other factors are not suitable for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-02-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Changes of quality of life (QoL) at 1 year after randomization compared with baseline | from randomization (day 1) up to 1 year
  The European Cancer Research and Treatment Collaboration (EORTC) Core Quality of Life Questionnaire (QLQ-C30) was used to assess patients' quality of life at 1 year after randomization (day 1). Proportion of improved/stable patients was considered as prespecified main endpoint. Improvement: at least 10 points improvement in Global Health status; Deterioration: Global Health status (Items 29 and 30 standardized score in QLQ-C30) decreased by at least 10 points; Other conditions are stable. Scoring method: In order to make the scores can be compared with each other, the range method is further adopted to carry out linear transformation, the Score for the field (RS,Raw Score) is obtained by adding up the Score of the items included in each field and dividing by the number of items included, and the crude scores are converted into standardized scores within 0-100.

SECONDARY OUTCOMES:
2-year survival rate | 2 year
  The probability of survival for 2 years from randomization. The patient's death for any cause is regarded as an end-point event. The time of death was recorded as the end event time. If no death was observed during the follow-up period, the date of the last confirmed survival was used as the time of deletion
Absolute changes of quality of life (QoL) compared with baseline | from randomization (day 1) up to two year
  The European Cancer Research and Treatment Collaboration Quality of Life Questionnaire-Colorectal Cancer 29 (EORTC QLQ-CR29). Standardized scores within 0-100. Describe the change in score.
Progression-free survival (PFS) | 2 year
  The time from randomization to the first occurrence of disease progression or death from all causes (whichever occurs first). If disease progression and death were not observed during follow-up, the date of the last tumor evaluation was used as the deletion time of PFS.
Performance Status score at first disease progression | from randomization (day 1) up to two year
  Zubrod-Eastern Cooperative Oncology Group(ECOG)-World Health Organization(WHO) was used to assess patients' performance status score for for patients with first disease progression after randomization. A minimum score of 0 is the best performance status; A maximum score of 5 is worst performance status.
Time to deterioration (TTD) | 2 year
  The time from randomization until patients reported the first deterioration (≥10 points from baseline) on each of the European Cancer Research and Treatment Collaboration (EORTC) Core Quality of Life Questionnaire(QLQ-C30) / The European Cancer Research and Treatment Collaboration Quality of Life Questionnaire-Colorectal Cancer 29 subscales (standardized scores within 0-100), and this was true for both consecutive evaluations, or for only one evaluation but death from any cause within the following 3 weeks.
Patient compliance | 2 year
  Patients who submit the electronic-Patient-Reported Outcomes questionnaire as required are considered to be completed
Patient satisfaction | 2 year
  Patients were followed up every 3 months for a satisfaction survey

OTHER OUTCOMES:
Accuracy of PRO to predict disease progression | 2 year
  To obtain a scale that can indicate disease progression of metastatic colorectal cancer and to determine the correlation coefficient between the item score of the scale and the degree of disease progression. A multi-item scale was put into this study, and the correlation between the items in the scale and disease progression was analyzed after the study.According to the correlation screening items, a scale was obtained to indicate the progression of metastatic colorectal cancer, and the correlation coefficient between the score of items in the scale and the degree of disease progression was calculated.The patient's disease progression will be determined by a combination of imaging and clinical symptoms
Economic assessment for ePRO compared to regular follow-up | 2 year
  the index for the incremental cost-effectiveness ratio (ICUR=ΔC/ΔQALY ), ePRO group patients compared to regular follow-up group patients, each for a unit of quality adjusted life years (QALY ), the extra cost

CONTACTS AND LOCATIONS:
Overall Officials: Yanqiao Zhang, Principal Investigator — Harbin Medical University Hospital
Locations (1):
- Harbin Medical University Hospital, Harbin, China